CLINICAL TRIAL: NCT02517372
Title: An Open-label, Single Center, Phase I, Dose Escalation Study Investigating the Safety, Tolerability and Pharmacokinetics of Pemirolast in Healthy Subjects
Brief Title: Study in Healthy Volunteers to Document Safety and Tolerability of Increasing Doses Pemirolast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RSPR Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: RSPR-PE-006
Record Dates: First submitted 2015-04-29; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pemirolast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohorte 1 (Active Comparator): "Low dose" pemirolast sodium (CRD007) given as one single dose on day 1, and thereafter twice daily for 3 days, followed by one single dose on day 5 and last day
  Interventions: Drug: CRD007
- Cohorte 2 (Active Comparator): "Medium dose" CRD007 given as one single dose on day 1, and thereafter twice daily for 3 days, followed by one single dose on day 5 and last day
  Interventions: Drug: CRD007
- Cohorte 3 (Active Comparator): "High dose" CRD007 given as one single dose on day 1, and thereafter twice daily for 3 days, followed by one single dose on day 5 and last day
  Interventions: Drug: CRD007

INTERVENTIONS:
Drug: CRD007
  Other Names: Pemirolast

SUMMARY:
This study is a single-centre, open-label, dose escalation , safety, tolerability and pharmacokinetics (PK) study in healthy male and female subjects. The study include a screening day and a 5-day dosing period. Subjects will be enrolled in sequential cohorts and each cohort will include 8 subjects. there will be 24 subjects total included in the study. The duration of the clinical part of the study will be approximately 2 months.

DETAILED DESCRIPTION:
Subjects meeting the eligibility criteria at screening will remain in the clinic from the evening preceding the first day of dosing (Day - 1) of the investigational medical product (IMP) and check out from the clinic 24 hours after the first dose administration of the IMP (in the morning of Day 2). Dose administration of the IMP in the evening of Day 2 and morning and evening dose for Days 3 and 4 will be performed at home. The subjects will check-in again in the morning of Day 5 and receive the last dose administration of the IMP and stay in the clinic 12 hours post dose. All subjects within the same cohort will receive the same dose of the IMP.

There will be 3 cohorts (dose-levels) with 8 subjects in each cohort corresponding to 24 subjects in total. Within a cohort the subjects will be dosed in groups of 4. There will be 24 hours between the dosing of the groups and 15 minutes between the dosing of the subjects in a group.

There will be an interval of approximately at least 1-week interval between the cohorts to allow time for compilation and evaluation of data for the Internal Safety Review Committee meeting.

Subsequent cohorts will be administered increasing doses until either the maximum tolerated dose (MTD) or the study maximum dose (SMD) has been reached.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, healthy subjects aged 19-65 years

Exclusion Criteria:

* Significant concurrent disease or medical conditions that are deemed to interfere with the safety or pharmacokinetics of CRD007 conduct of the trial

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Events as a measure of Safety and Tolerability | Change from baseline to day 5 (12 hours post dose)
Results of physical examination as a composite outcome measure of Safety and Tolerability | Change from baseline to day 5 (12 hours post dose)
ECG recording as a measure of Safety and Tolerability | Change from baseline to day 5 (12 hours post dose)
Vital signs (Blood Pressure and Pulse Rate) as a composite outcome measure of Safety and Tolerability | Change from baseline to day 5 (2 hours post dose)

SECONDARY OUTCOMES:
Composite outcome measure consisting of multiple pharmacokinetics measures (Area Under the plasma concentration-time Curve (AUC), Plasma elimination half-life (t½), Time to maximum plasma drug concentration (Tmax), and Peak Plasma Concentration (Cmax)) | Blood sampling day 1 up to 24 hrs post dose and day 5 up to 24 hrs post dose